CLINICAL TRIAL: NCT00747916
Title: A Pilot Study of the Safety, Efficacy, and Side Effects of Interventional Cryotherapy for the Eradication of Disease in the Pleural Space ("ICE PLS")
Brief Title: Safety, Efficacy, and Side Effects Study of Interventional Cryotherapy in the Pleural Space("ICE PLS")
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Business Reasons
Sponsor: CSA Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 17-00027
Record Dates: First submitted 2008-09-04; First posted 2008-09-08 (Estimated); Results first posted 2015-06-08 (Estimated); Last update posted 2015-07-16 (Estimated); Status verified 2015-06

CONDITIONS: Cancer; Pleural Neoplasms
Keywords: Parietal pleura; Neoplasms; Pleural Surface; Pleural Neoplasms; Lung Cancer
MeSH Terms: conditions — Neoplasms; Pleural Neoplasms; Lung Neoplasms | interventions — Drug Delivery Systems; Cryotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- CryoSpray Ablation (TM) System (Experimental): subjects will receive cryotherapy using the CryoSpray Ablation (TM) System DOSE: up to 3 cycles of 10-40 second sprays
  Interventions: Device: CryoSpray Ablation (TM) System

INTERVENTIONS:
Device: CryoSpray Ablation (TM) System — Subjects will be treated with spray cryotherapy using the CryoSpray Ablation (TM) System at Day 0 using up to 3 cycles of 10-40 second sprays as the studied dosimetry and will cover the affected area, including the tumor and the parietal pleural surface. If disease exists bilaterally, only one side will be sprayed. Subjects will be assessed 2-5 days from the initial treatment (Day 0) to check for mucosal sloughing, to reassess tumor burden and for additional CSA therapy as needed.
  Other Names: CSA (TM) System; CryoSpray Therapy; CSA; Cryotherapy; Cryospray

SUMMARY:
The purpose of this study is to evaluate the safety, efficacy, and side effects of the CryoSpray Ablation(TM) System (CSA(TM) System) to treat neoplastic lesions on the parietal pleural surface.

DETAILED DESCRIPTION:
The proposed study is a pilot study consisting of an estimated 10 subjects with biopsy-proven metastatic cancer in the parietal pleural surface treated with CryoSpray at dye marked metastatic foci.

Initial treatment dosimetry will be up to 3 cycles of 10-40 second sprays. If necessary, dosimetry changes may occur after 3 subjects are treated and observed. It is unknown if dosimetry will need to be increased to enhance effectiveness. The PI may increase dosimetry by 1 cycle after each subject is treated and observed as a conservative approach to efficacy determination. If disease exists bilaterally, only one side will be sprayed.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age
* Deemed a candidate for cryotherapy based on physician physical or medical history review
* Deemed operable based on institutional criteria
* Able to sign informed consent
* Documented lung or other visceral cancer with pleural involvement.
* WBC > 4,000/mm3, platelets >100,000mm3
* Physically well enough to undergo moderate sedation and pleuroscopy
* Female patients must be HCG negative
* There should be direct evidence of disease progression despite treatment in previously treated patients

Exclusion Criteria:

* Pregnant or nursing
* Planning to sire a child while enrolled in the study
* Known history of unresolved drug or alcohol dependency that would limit ability to comprehend or follow instructions related to informed consent, post-treatment instructions, or follow-up guidelines.
* Refusal or inability to give consent.
* Concurrent chemotherapy.
* Medical contraindication or potential problem that would preclude study participation
* Concurrent participation in other experimental studies
* Uncontrolled coagulopathy or bleeding diathesis
* Serious medical illness, including:
* Uncontrolled congestive heart failure
* Uncontrolled angina
* Myocardial infarction
* Cerebrovascular accident within 6 months prior to study entry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2008-08; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gordon Downie, M.D., Ph.D, Principal Investigator — University of Texas Health Center at Tyler
Locations (1):
- University of Texas Health Center at Tyler - Titus Regional Hospital, Tyler, Texas, United States

REFERENCES:
- [Background] Johnston MH, Eastone JA, Horwhat JD, Cartledge J, Mathews JS, Foggy JR. Cryoablation of Barrett's esophagus: a pilot study. Gastrointest Endosc. 2005 Dec;62(6):842-8. doi: 10.1016/j.gie.2005.05.008. PMID 16301023
- [Background] Johnston CM, Schoenfeld LP, Mysore JV, Dubois A. Endoscopic spray cryotherapy: a new technique for mucosal ablation in the esophagus. Gastrointest Endosc. 1999 Jul;50(1):86-92. doi: 10.1016/s0016-5107(99)70352-4. PMID 10385730
- [Background] Ell C, May A, Gossner L, Pech O, Gunter E, Mayer G, Henrich R, Vieth M, Muller H, Seitz G, Stolte M. Endoscopic mucosal resection of early cancer and high-grade dysplasia in Barrett's esophagus. Gastroenterology. 2000 Apr;118(4):670-7. doi: 10.1016/s0016-5085(00)70136-3. PMID 10734018
- [Background] Champion G, Richter JE, Vaezi MF, Singh S, Alexander R. Duodenogastroesophageal reflux: relationship to pH and importance in Barrett's esophagus. Gastroenterology. 1994 Sep;107(3):747-54. doi: 10.1016/0016-5085(94)90123-6. PMID 8076761
- [Background] Eisen GM, Sandler RS, Murray S, Gottfried M. The relationship between gastroesophageal reflux disease and its complications with Barrett's esophagus. Am J Gastroenterol. 1997 Jan;92(1):27-31. PMID 8995932
- [Background] Johnston MH. Cryotherapy and other newer techniques. Gastrointest Endosc Clin N Am. 2003 Jul;13(3):491-504. doi: 10.1016/s1052-5157(03)00044-8. PMID 14629105
- [Background] Cash BD, Johnston LR, Johnston MH. Cryospray ablation (CSA) in the palliative treatment of squamous cell carcinoma of the esophagus. World J Surg Oncol. 2007 Mar 16;5:34. doi: 10.1186/1477-7819-5-34. PMID 17367523
- [Background] Field JK, Youngson JH. The Liverpool Lung Project: a molecular epidemiological study of early lung cancer detection. Eur Respir J. 2002 Aug;20(2):464-79. doi: 10.1183/09031936.02.00290202. PMID 12212983
- [Background] Pinsonneault C, Fortier J, Donati F. Tracheal resection and reconstruction. Can J Anaesth. 1999 May;46(5 Pt 1):439-55. doi: 10.1007/BF03012943. PMID 10349923
- [Background] Dumot JA. Cryotherapy Ablation for Esophageal HGD or IMCA in High Risk, Non-Surgical Patients. DDW2007 Abstract submission. Cleveland Clinic Foundation (pending publication)
- [Background] Greenwald BD. CryoSpray Ablation of Early Esophageal Cancer. DDW 2007 Abstract submission. University of Maryland Medical Center. (pending publication)
- [Background] Johnston M, Horwhat J, Dubois A, Schoenfeld P. Endoscopic cryotherapy in the swine esophagus: A follow-up study (Abstract). Gastrointestinal Endoscopy 49:AB126, 1999.
- [Background] Johnston MH, Horwhat JD, Haluska, Moses FM. Depth of injury following endoscopic spray cryotherapy: EUS assisted evaluation of mucosal ablation and subsequent healing in the swine model (Abstract). Gastrointestinal Endoscopy 51: AB98, 3462, 2000.
- [Background] Johnston MH. Endoscopic cryotherapy: A new ice age in gastroenterology? Medscape Gastroenterology 2: 187, 2000.
- [Background] Eastone JA, Horwhat D, Haluska O, Mathews J, Johnston M. Cryoablation of swine esophageal mucosa: A direct comparison to argon plasma coagulation (APC) and multipolar electrocoagulation (MPEC) [Abstract] Gastrointestinal Endoscopy 53: A3448, 2001.
- [Background] Johnston MH, Eastone JA, Horwhat JD. Reversal of Barrett's esophagus with cryotherapy [Abstract]. American Journal of Gastroenterology 98(9 Suppl): A30, S11, 2003.
- [Background] Johnston MH, Cash BD, Horwhat JD, Johnston LR, Dykes CA, Mays HS. Cryoablation of Barrett's Esophagus (BE) [Abstract]. Gastroenterology 130 (4, Suppl.2): A640, 2006.
- [Background] Johnston MH, Cash BD, Dykes CA, Mays HS, Johnston LR. Cryoablation of dysplasia in Barrett's Esophagus (BE) and early stage esophageal cancer [Abstract]. Gastrointestinal Endoscopy 63 (5): April, 2006.

RESULTS

PARTICIPANT FLOW:
Groups:
- All Participants ICE PLS: The study consists of one arm. All subjects enrolled in All participants ICE PLS
Period: Overall Study
Arm/Group | All Participants ICE PLS
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | All Participants ICE PLS
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 1
Age, Continuous [Mean (Full Range); unit: years] | 59 [49 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: To Reduce Tumor Burden in the Pleural Space, as Determined by Visual Inspection and Biopsy of the Treatment Sites 2-5 Days Post Treatment. Safety Endpoint Clinical and Radiographic Status at 30 Days Post CryoSpray Treatment and Adverse Events.
Time Frame: 1 year
Population: zero participants analyzed due to early termination of study
Arm/Group | All Participants ICE PLS
Number analyzed (Participants) | 0

2. Secondary Outcome: To Determine if CryoSpray Causes a Pleurodesis Effect. To Determine if CryoSpray Affects Production of Malignant Effusion Within the Treated Pleural Cavity. To Determine if Pleural Cavity Treatment With CryoSpray is Dosimetry Dependent.
Time Frame: 1 year
Population: zero participants analyzed due to early termination of study
Arm/Group | All Participants ICE PLS
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | All Participants ICE PLS
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No